CLINICAL TRIAL: NCT05961397
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Pharmacokinetics of CIN-107 in Subjects With Varying Degrees of Hepatic Function
Brief Title: Phase 1 PK Study to Evaluate the PK of CIN-107 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-115
Record Dates: First submitted 2023-07-03; First posted 2023-07-27 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: hepatic impairment; PK; baxdrostat
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal hepatic function group (Experimental): Subjects with normal hepatic function
  Interventions: Drug: baxdrostat
- Moderate hepatic impairment group (Experimental): Subjects with a Child-Pugh score of 7 to 9 (Category B) at screening
  Interventions: Drug: baxdrostat

INTERVENTIONS:
Drug: baxdrostat — single oral dose of baxdrostat 10 mg
  Other Names: CIN-107

SUMMARY:
The goal of this Phase 1, open-label, single-dose, parallel-group study is to evaluate the pharmacokinetics (PK) of a single 10-mg oral dose of baxdrostat in subjects with varying degrees of hepatic function. The main objectives are to:

* To assess the safety and tolerability of baxdrostat following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function; and
* To characterize the PK of baxdrostat following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function.

Participants were administered a single 10-mg oral dose of baxdrostat in the fasted state the morning of Day 1. Plasma samples were drawn at various timepoints. Safety assessments included adverse events, vital signs, 12-lead electrocardiograms (ECGs), clinical laboratory evaluations, and physical examinations.

Twenty subjects in 2 groups based on the Child-Pugh classification in the protocol at screening: up to 10 subjects in the normal hepatic function group and up to 10 subjects in the moderate hepatic impairment group. Twenty subjects entered and completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 80 years, inclusive, and in stable health condition. (For hepatically impaired subjects, their hepatic function category must be stable for a minimum of 3 months prior to screening.)
* Is a non-nicotine user or smokes =<10 cigarettes/day;
* Has a BMI between 18 and 42 kg/m2, inclusive;
* Is able to understand and willing to comply with study procedures and restrictions and provide written informed consent;
* if a male subject with a female partner of childbearing potential must agree to use 2 medically accepted, highly effective methods of birth control for 90 days.
* if male, must agree to abstain from sperm donation for 90 days; and
* if female with a male partner, must be surgically sterile, postmenopausal, or agree to use 2 medically accepted, highly effective methods of birth control from Day -14 until 60 days after study drug dosing

Main Exclusion Criteria:

* Personal or family history of long QT syndrome, torsades de pointes, or other complex ventricular arrhythmias, or family history of sudden death;
* History of, or current, clinically significant arrhythmias;
* Prolonged QTcF (>460 msec) based on the average of triplicate ECGs;
* Estimated glomerular filtration rate (or creatinine clearance) <50 mL/min/1.73 m2;
* Evidence of any of the following: Encephalopathy grade 2 or worse, Seated systolic BP >160 mmHg and/or diastolic BP >100 mmHg, or systolic BP <90 mmHg and/or diastolic BP <50 mmHg, resting heart rate >100 beats per minute (bpm) or <50 bpm, Oral temperature >37.6°C (>99.68°F), Respiration rate <12 or >20 breaths per minute, symptomatic postural tachycardia or orthostatic hypotension, abnormal serum potassium >upper limit of normal range, abnormal serum sodium <130 mEq/L, positive test for HIV antibody, hepatitis C , hepatitis B , or SARS-CoV-2 RNA
* Current treatment with weight loss medication or prior weight loss surgery;
* Use of a moderate or strong inhibitor of CYP3A4 within 14 days prior to the dose of study drug OR use of a moderate or strong inducer of CYP3A4 within 28 days prior to the dose of study drug;
* Corticosteroid use (systemic or extensive topical use) within 3 months prior to study drug dosing
* Pregnant, breastfeeding, or planning to become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function. | up to 72 hours post-dose
  The safety and tolerability of baxdrostat was assessed throughout the study based on incidence of treatment emergent adverse events (AEs), following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function.
Area under the curve (AUC) for baxdrostat and the CIN-107-M metabolite following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function | up to 72 hours post-dose
  Measurement of plasma concentrations of baxdrostat and its major metabolite CIN-107-M. AUC [0 to 24 hours, 0 to last quantifiable concentration, and 0 to infinity of baxdrostat] will be determined for baxdrostat and the CIN-107M metabolite.
Maximum Plasma Concentration [Cmax] of baxdrostat and the CIN-107-M metabolite following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function. | up to 72 hours post-dose
  Cmax will be determined for baxdrostat and the CIN-107M metabolite
Time to Maximum Plasma Concentration [Tmax] of baxdrostat and the CIN-107-M metabolite following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function. | up to 72 hours post-dose
  Tmax will be determined for baxdrostat and the CIN-107M metabolite
Terminal elimination half-life of baxdrostat and the CIN-107-M metabolite following administration of a single oral dose of baxdrostat to subjects with varying degrees of hepatic function. | up to 72 hours post-dose
  Terminal elimination half-life will be determined for baxdrostat and the CIN-107M metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Cruz, MD, Principal Investigator — Advanced Pharma CR; William B Smith,, MD, Principal Investigator — Alliance for Multispecialty Research; Zeid Kayali, MD, Principal Investigator — Inland Empire Clinical Trials; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Eric Lawitz, MD, Principal Investigator — American Research Corporation at the Texas Liver Institute
Locations (5):
- United States (5):
  - Inland Empire Clinical Trials, Rialto, California
  - Advanced Pharma CR, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, Knoxville, Tennessee
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-115&attachmentIdentifier=39073201-1e04-4750-aff3-5f7739890c35&fileName=cin-107-115-csr-synopsis_Redacted.pdf&versionIdentifier=